CLINICAL TRIAL: NCT06306300
Title: Randomized Open-label and Non-inferiority Clinical Trial to Evaluate the Safety, Adherence, and Cost-effectiveness of Simplified and Decentralized Hepatitis C Treatment in Primary Health Care Compared to Standard-of-care in the Brazilian Public Health System
Brief Title: Safety and Efficacy of Decentralized HCV Treatment vs Standard-of-Care in Rio de Janeiro (Brazil)
Acronym: HCVPCL05/20
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Hugo Perazzo Pedroso Barbosa, Principal Investigator, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 445957/2020-4
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; Primary health care; Hepatitis C virus self-test
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Study I is a population-based cross-sectional screening study (n=30,000 individuals) to determine the prevalence of HCV infection in people attending a Basic Health Care Unit. The sub-study associated with Study I is a cross-sectional study to assess the usability of a self-test for the detection of HCV antibodies in oral fluid (n=1,500 participants included in Study I). Study II is a phase IV open-label randomized clinical trial (1:1) to evaluate the non-inferiority of simplified and decentralized hepatitis C treatment ("Simplified-and-Decentralized (SD) HCV treatment"; experimental arm) compared to specialist reference treatment ("Standard-of-Care (SC) HCV treatment"; control arm) within the SUS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study I (No Intervention): Study I is a population-based cross-sectional screening study (n=30,000 individuals) using rapid tests to determine the prevalence of HCV infection in people attending a Basic Health Care Unit.
- Substudy I (No Intervention): The sub-study associated with Study I is a cross-sectional study to assess the usability of a self-test for the detection of HCV antibodies in oral fluid (n=1,500 participants included in Study I).
- Study II - Specialist (Active Comparator): HCV standard-of-care treatment"; control arm. Participants randomized for the Standard-of-Care HCV treatment arm will be referred for the usual treatment of hepatitis C by specialists (hepatologists and/or infectious disease specialists) at a tertiary center [INI/FIOCRUZ or Hospital Universitário Clementino Fraga Filho (HUCFF/UFRJ)]. Participants will be treated with the pan-genotypic therapeutic regimen "single-pill daily," at a fixed dose and duration: sofosbuvir/velpatasvir 400/100 mg (Epclusa, Gilead Sciences, USA) 1 tablet orally per day for 12 weeks.
  Interventions: Drug: Specialist - Epclusa 400Mg-100Mg Tablet
- Study II - Non Specialist (Active Comparator): Decentralized hepatitis C treatment ("DS HCV treatment"; experimental arm).Participants randomized for the "Decentralized-and-Simplified HCV treatment" (DS HCV treatment) arm will be referred for simplified treatment of chronic hepatitis C at the Primary Health Care unit where participants were included in Study I and are registered for care. The treatment will be conducted by a non-specialist physician (general practitioner or family doctor) after training provided by a specialist (hepatologist) on the treatment of patients with hepatitis C using DAAs. Participants will be treated with a pan-genotypic therapeutic regimen, a fixed-dose, single-pill daily: sofosbuvir/velpatasvir 400/100 mg (Epclusa, Gilead Sciences, USA), 1 tablet orally per day for 12 weeks.
  Interventions: Drug: Non- specialist - Epclusa 400Mg-100Mg Tablet

INTERVENTIONS:
Drug: Specialist - Epclusa 400Mg-100Mg Tablet — HCV-positive participants from study 1 will be randomized to be treated in the specialist arm, which consists of follow-up by a specialized doctor.
  Other Names: Standard-of-Care (SC) HCV treatment
  Arms: Study II - Specialist
Drug: Non- specialist - Epclusa 400Mg-100Mg Tablet — HCV-positive participants from study 1 will be randomized to be treated in the specialist arm, which consists of follow-up by non-specialized doctor.
  Other Names: Simplified-and-Decentralized (SD) HCV treatment
  Arms: Study II - Non Specialist

SUMMARY:
Up to 650,000 people in Brazil are living with chronic hepatitis c virus (HCV) infection. Hepatitis C is a silent disease, and up to 20% of cases can progress to liver cirrhosis and its complications. Rapid tests for diagnosis of HCV infection and non-invasive methods for detecting liver cirrhosis are available in the Brazilian Public Health System. Additionally, safe and highly effective drugs (direct-acting antivirals, DAAs) have been delivered for free for hepatitis C treatment by the Brazilian Unified Health System (Sistema Único de Saúde, SUS) since 2015. Sustained virological response (SVR) rates with DAAs in studies conducted in Brazil and Latin America were higher than 90%. Despite the availability of rapid tests for early diagnosis and effective drugs, the HCV continuum of care remains deficient in Brazil. It is estimated that only 10% of individuals known to have hepatitis C achieve HCV cure (SVR). This is explained by multiple barriers from diagnosis to treatment access, such as low rates of population screening (HCVST are not available in Brazil) and few available slots in tertiary centers for hepatitis C treatment by specialists. International studies have described that SVR rates by simplified hepatitis C treatment performed by non-specialists in the Primary Care System were similar to those treated in tertiary centers by specialists (standard-of-care). However, the optimal strategy for managing hepatitis C within the Brazilian-SUS remains unclear.This project aims to evaluate the improve of the HCV continuum of care by a implementation of a test-and-treat strategy in the Primary Care System in Brazil. The project consists of two parallel studies (and a sub-study).

The project consists of two parallel studies (and a sub-study). Study I is a population-based cross-sectional screening study using rapid tests to determine the prevalence of HCV infection in people attending a Basic Health Care Unit. The sub-study associated with Study I is a cross-sectional study to assess the usability of a self-test for the detection of HCV antibodies in oral fluid (participants included in Study I). Study II is a phase IV open-label randomized clinical trial to evaluate the non-inferiority of simplified and decentralized hepatitis C treatment ("Simplified-and-Decentralized (SD) HCV treatment"; experimental arm) compared to specialist reference treatment ("Standard-of-Care (SC) HCV treatment"; control arm) within the SUS.

DETAILED DESCRIPTION:
In Brazil, liver cirrhosis was the cause of death for over 265,000 people between 2000 and 2012. The mortality rate from cirrhosis in 2012 was 12 deaths per 100,000 inhabitants, and the number of deaths from liver cirrhosis increased by about 22% in the last decade.

Recently, hepatitis C treatment has been revolutionized by the use of direct-acting antivirals (DAAs), which are safe and highly effective oral medications. Cure rates for hepatitis C, known as sustained virological response (SVR), in studies conducted in Brazil and Latin America were higher than 90%. Hepatitis C cure (SVR) is associated with a reduction in the incidence of HCC, the need for liver transplantation, improvement in quality of life, and a decrease in HCV transmission. These new medications have been available for hepatitis C treatment through the Brazilian Public Health System, known as Sistema Único de Saúde (SUS) since 2015.

The Ministry of Health of Brazil signed an agreement with the WHO in 2016 and with the goal of defining public health strategies to eliminate viral hepatitis by 2030, reducing new infections by 90% and global hepatitis-related mortality by 65%.

Identifying individuals with HCV infection is crucial for the (micro) elimination of hepatitis C. The majority of chronically infected HCV patients are asymptomatic until the development of liver cirrhosis and/or its complications. Therefore, screening for HCV infection should be performed in individuals, even when asymptomatic, through HCV antibody (HCVab) test. Currently, HCV rapid tests (HCVRT) in fingerstick blood with results in 15-20 minutes are available in Brazil.

Historically, HCV screening was recommended for individuals over 40 years of age and high-risk populations for HCV infection, such as people who inject drugs (PWID), prisoners, and men who have sex with men (MSM). However, recent international guidelines recommend screening for all individuals aged 18-79. Active HCV infection should be confirmed by detecting HCV viral load using molecular tests by polymerase chain reaction (PCR). Currently, the identification of HCV-RNA by PCR as a point-of-care tests (PoCT), GeneXpert® System, is also possible. The Xpert HCV VL Fingerstick test has excellent accuracy for detecting HCV-RNA in fingerstick blood, providing results in up to 105 minutes.. Liver elastography is a rapid imaging method (< 5 minutes), similar to abdominal ultrasound, painless, and free of complications, that can be performed at the bedside and provides real-time results for fibrosis stage/liver cirrhosis diagnosis. The technical principle of this method is based on measuring the propagation of ultrasound waves, called shear waves, through the liver parenchyma, estimating the organ's fibrosis degree through liver stiffness measurement (LSM). Currently, portable/semi-portable hepatic elastography devices are available, allowing for the staging of liver fibrosis in regions with difficult access to healthcare.

Globally, the HCV continuum of care is still deficient, as only about 10% of identified hepatitis C patients achieve SVR. Brazil also observes a similar scenario of deficiencies in the HCV cascade of care. People living with HCV are typically treated in tertiary centers by specialists (infectious disease specialists, hepatologists, gastroenterologists). Multiple pre-treatment visits (diagnostic confirmation, biological analyses, and staging of liver fibrosis) are required, along with visits during treatment (clinical visits and biological analyses) and after medication use (evaluation of hepatitis C cure). This process can be even more complicated in certain stigmatized, highly vulnerable populations, and/or those with difficult access to healthcare. The hepatitis C treatment cascade can be improved, especially with recent advances in techniques for diagnosing/confirming HCV infection and the availability of pan-genotypic and simple therapeutic regimens (one tablet orally per day for 12 weeks, "one-size-fits-all"), extremely safe and highly effective (even in patients with advanced fibrosis/liver cirrhosis). The simplification of hepatitis C treatment leads to higher detection and treatment rates (increased access to treatment), rapid initiation of treatment post-diagnosis (rapid linkage-to-care), reduced HCV transmission (treatment as a prevention tool), and cost reduction associated with cirrhosis complications/liver transplantation. Additionally, international studies have described that the response rates to hepatitis C treatment by non-specialists in the Primary Health Care System with DAAs seems to be similar to those treated by specialists. However, the best strategy for managing hepatitis C within the Brazilian-SUS is not yet widely defined.

ELIGIBILITY:
Study I and Sub-Study

Inclusion Criteria:

- Age between 18-79 years-old

Exclusion Criteria:

* Presence of a disease that need urgent/emergency treatment and/or acute febrile illness, such as COVID-19, Dengue, Zyca virus infection or Chikungunya
* Lack of capacity to sign the informed consent or refuse to participate

Study II

Inclusion Criteria:

* Age between 18 and 79 years old.
* Presence of active/chronic hepatitis C, defined by a positive HCVab test and detectable HCV-RNA

Exclusion Criteria:

* Children and adolescents (< 18 years old)
* Pregnancy, defined by a positive β-HCG urinary test
* Lactating individuals
* Co-infection with HBV or HIV
* Regular use of medications with potential drug interactions or contraindication for co-administration with SOF/VEL
* Presence of severe acute illness, active neoplasia, solid organ transplant, or use of immunosuppressive medications
* Presence of clinical signs of decompensated liver cirrhosis (ascites, hepatic encephalopathy, report of a recent episode of gastrointestinal bleeding within the last 12 weeks)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HCV infection | 1 month
  The primary outcome of Study I will be the assessment of the prevalence of HCV infection in users of the Felippe Cardoso Family Clinic, Zilda Arns Family Clinic, and/or Klebel de Oliveira Rocha Family Clinic, located in the municipality of Rio de Janeiro.
The effectiveness of the HCV treatment with test results. | 1 month
  The primary outcome of Study II will be the effectiveness of the HCV treatment in both arms, translated by sustained virological response (SVR12), characterized by undetectable HCV-RNA by the PCR method at least 12 weeks after the end of treatment with SOF/VEL. Comparison of test results at the beginning and end of treatment
Usability of the result of a self-test HCV | 1 month
  Evaluate the interpretability of the result of a self-test for the detection of HCV antibodies (HCVab) in oral fluid in a subset of participants included in Study I (adults performing HCV testing). Comparison of the results of the tests carried out by the participant with those of the professional.

SECONDARY OUTCOMES:
Proportion between positive and negative | 1 month
  Proportion of individuals with positive HCV anti-body (HCVab) test and undetectable HCV-RNA (spontaneous HCV clearance or false negative HCV ab test)
Participants with fibrosis/cirrhosis | 1 month
  Prevalence of advanced liver fibrosis/cirrhosis (hepatic elastography ≥ 9.5 kPa) in people with chronic hepatitis C (reactive HCVab test & detectable HCV-RNA).
Participants who denied the treatment | 1 month
  Proportion of patients who refuse treatment for chronic hepatitis C.
cost per detected participant | 1 month
  Cost per case detected with HCV infection
Unscheduled visits during treatment | 3 months
  Rate of unplanned clinical visits during HCV treatment (from Day 0 to Week 12)
Improvement of liver fibrosis stage | 1 year
  Change in liver fibrosis stage, measured by hepatic elastography between the entry study assessment (Day 0) and the end-of-study assessment (Week 36 ± 12) among participants with SVR.
Quality of life data | 1 month
  Quality of life (health-related utility) before and after HCV cure (SVR).
Cost of treatment for participant | 1 month
  Cost per case who achieved SVR
Adherence to treatment | 1 month
  Adherence to SOF/VEL treatment measured by attendance at scheduled visits and reported by participants

OTHER OUTCOMES:
Participant´s Ability to use the test | 1 month
  Assess the ability to perform the oral fluid HCV self-test
Participant preference for types of tests | 1 month
  The participant's information will be collected in the questionnaire, which will contain data on their preference between the two types of tests HCV self-testing using oral fluid and the conventional rapid test (fingerstick blood sample performed by a healthcare professional) .
Participant understanding to interpret his result | 1 month
  By comparing the results of the tests carried out by the participant and the health professional, it will be identified whether the participant performed the correct reading.
Test Performance | 1 month
  By comparing the results of the tests carried out by the participant and the health professional, it will be identified whether the participant performed the test correctly.
Test Accuracy | 1 month
  Comparison of the results of the self-test for HCV in oral fluid (self-testing and performed by a healthcare professional) compared to the conventional rapid test, whether they have the same precision of results. .

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Evandro Chagas National Institute of Infectious Diseases, Rio de Janeiro, Rio de Janeiro/RJ
  - Hugo Perazzo, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No
There is a confidentiality of participant data.